CLINICAL TRIAL: NCT01685125
Title: A Randomized Phase II Trial of Dasatinib Plus Abiraterone Compared to Abiraterone Alone for Metastatic, Castration-Resistant Prostate Cancer Prior to Chemotherapy
Brief Title: Abiraterone Acetate and Prednisone With or Without Dasatinib in Treating Patients With Metastatic Hormone-Resistant Prostate Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4P-12-1; NCI-2012-01485 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-09-11; First posted 2012-09-13 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-06

CONDITIONS: Hormone-resistant Prostate Cancer; Recurrent Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Dasatinib; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (abiraterone acetate, prednisone) (Active Comparator): Abiraterone acetate 1000 mg PO QD and Prednisone 5 mg PO BID on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: abiraterone acetate; Drug: prednisone
- Arm B (abiraterone acetate, prednisone, dasatinib) (Experimental): Abiraterone acetate 1000 mg PO QD, Prednisone 5 mg PO BID, and dasatinib 100 mg PO QD on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: abiraterone acetate; Drug: dasatinib; Drug: prednisone

INTERVENTIONS:
Drug: abiraterone acetate — Given PO
  Other Names: CB7630; Zytiga
Drug: dasatinib — Given PO
  Other Names: BMS-354825; Sprycel
  Arms: Arm B (abiraterone acetate, prednisone, dasatinib)
Drug: prednisone — Given PO
  Other Names: DeCortin; Deltra

SUMMARY:
This phase II trial studies how well giving abiraterone acetate and prednisone with or without dasatinib works in treating patients with metastatic, hormone-resistant prostate cancer. Androgens can cause the growth of prostate cancer cells. Antihormone therapy, such as abiraterone acetate, may lessen the amount of androgens made by the body. Dasatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether abiraterone acetate and prednisone is more effective than abiraterone acetate, prednisone, and dasatinib in treating prostate cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the progression-free survival of men with metastatic castration-resistant prostate cancer treated with abiraterone (abiraterone acetate) plus dasatinib to that of men treated with abiraterone alone.

SECONDARY OBJECTIVES:

I. To describe the toxicity profile of the combination, as well as the rate of prostate-specific antigen (PSA) response, objective responses, and changes in circulating tumor cell (CTC) numbers.

OUTLINE: Patients are randomized to 1 of 2 treatment arms. ARM A: Patients receive abiraterone acetate 1000 mg orally (PO) once daily (QD) and prednisone 5 mg PO twice daily (BID) on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive abiraterone acetate and prednisone as patients in arm A. Patients also receive dasatinib 100 mg PO QD on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic, castration-resistant prostate cancer

  * Defined as evaluable radiographic disease with rising PSA x 2 (at least 1 week apart) or radiographic progression (new soft tissue/bone lesions or enlarging soft tissue lesions) despite medical or surgical castration
  * No limit on prior hormonal therapies (i.e. anti-androgens, ketoconazole) except that subject must not have received abiraterone previously
  * No limit on prior biologic therapies (i.e. immune therapy, antiangiogenic, targeted) except that patient should not have received dasatinib or other v-src sarcoma (Schmidt-Ruppin A-2) viral oncogene homolog (avian) (src)-targeted therapy
* No prior chemotherapy for metastatic disease

  * Subjects who have received chemotherapy in the neoadjuvant or adjuvant setting will be eligible provided chemotherapy was completed > 6 months prior to enrollment
* Eastern Cooperative Oncology Group (ECOG) 0-2
* Total bilirubin =< 1.5 times the institutional upper limit of normal (ULN) except for Gilbert's syndrome
* Hepatic enzymes (aspartate aminotransferase [AST], alanine aminotransferase [ALT] ) =< 2.5 times the institutional ULN
* Serum sodium (Na), potassium (K+), magnesium (Mg+), phosphate and calcium (Ca+) > lower limit of normal (LLN)
* Serum creatinine =< 1.5 time the institutional ULN
* Hemoglobin (Hb) >= 9
* Platelets >= 100,000
* Absolute neutrophil count (ANC) >= 1000
* Ability to take oral medication (study medications must be swallowed whole)
* Men with fathering potential must agree to use contraception throughout study treatment; acceptable methods include: condoms, sponge, intrauterine device (IUD), oral contraceptives
* Concomitant medications * Patient agrees to discontinue St. Johns wort while receiving dasatinib therapy (discontinue St. Johns wort at least 5 days before starting dasatinib)

Exclusion Criteria:

* Known hepatitis B or C or human immunodeficiency virus (HIV), regardless of viral load

  * Testing for the purposes of enrollment is not mandatory, however a documented history of these infections will be exclusionary due to concerns for drug-drug interactions with antivirals and potential for increased risk of liver toxicity
* Radiation for palliation of bony metastases within the preceding 2 weeks
* Prior chemotherapy for metastatic castration-resistant prostate cancer (CRPC)

  * Immune therapy with sipuleucel-T is allowed, provided the last infusion was >= 28 days prior to study therapy and there has been at least one documented PSA value rising after completion of sipuleucel-T therapy or progression of disease on imaging after sipuleucel-T
* Malignancy (aside from prostate cancer) which required radiotherapy or systemic treatment within the past 5 years

  * Superficial bladder cancer treated with intravesical therapy and currently in remission will not be an exclusion
  * Skin cancers will not be an exclusion, except for melanoma with a thickness > 1 mm
* Concurrent medical condition which may increase the risk of toxicity, including:

  * Pleural or pericardial effusion of any grade at the time of study entry
  * Cardiac symptoms; any of the following should be considered for exclusion: ** Uncontrolled angina, congestive heart failure or myocardial infarction (MI) within (6 months)

    * Diagnosed congenital long QT syndrome
    * Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes) ** Prolonged QTc/f interval on pre-entry electrocardiogram (> 450 msec)
    * Hypokalemia or hypomagnesemia if it cannot be corrected prior to abiraterone administration
* History of significant bleeding disorder unrelated to cancer, including:

  * Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease)
  * Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies)
  * Ongoing or recent (=< 3 months) significant gastrointestinal bleeding
* Prohibited treatments and/or therapies

  * Should not be on any additional anti-cancer therapy except for luteinizing hormone-releasing hormone (LHRH) agonist/antagonist; specifically excluded medications include ketoconazole, estrogens, and anti-androgens
  * Category I drugs that are generally accepted to have a risk of causing Torsades de pointes including: (Patients must discontinue drug 7 days prior to starting dasatinib)

    * Quinidine, procainamide, disopyramide
    * Amiodarone, sotalol, ibutilide, dofetilide
    * Erythromycin, clarithromycin
    * Chlorpromazine, haloperidol, mesoridazine, thioridazine, pimozide
    * Cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine
* Prisoners or subjects who are involuntarily incarcerated
* Subjects who are compulsorily detained for treatment of either a psychiatric or physical (eg, infectious disease) illness

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2012-09; Primary Completion 2016-03 (Actual); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From the start of abiraterone acetate until first evidence of disease progression or until death from any cause, whichever occurs first, assessed up to 3 years
  PFS defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. A one-sided, 0.05-level log rank test will be used to compare the two arms in terms of PFS. PFS will be estimated using the product-limit method of Kaplan and Meier.

SECONDARY OUTCOMES:
Overall response | Up to 3 years
  Overall response defined as the percent of subjects whose best response is a complete response or partial response based on RECIST version 1.1. Exact 95% confidence intervals will be calculated for this estimate.
PSA change response according to PSA Working Group Criteria 2 | Baseline and 12 weeks
  PSA changes will be summarized for each arm also using waterfall plots as well as standard descriptive statistics.
Overall survival | From start of abiraterone acetate and/or dasatinib treatment until death due to any cause or time the patient was last known to be alive, assessed up to 3 years
  Estimated using the product-limit method of Kaplan and Meier. The probability of remaining alive at 6, 12, 18 and 24 months, with the associated Greenwood's standard errors, will be summarized.
Intent-to-treat analysis | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Dorff, Principal Investigator — University of Southern California
Locations (1):
- USC Norris Comprehensive Cancer Center, Los Angeles, California, United States